CLINICAL TRIAL: NCT02557880
Title: Does the Utilization of a Sleep Application Diary Improve Sleep Hygiene in Adolescents?
Brief Title: Sleep Application Diary and Sleep Hygiene in Adolescents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not get teenagers to enroll
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Cheryl Tierney, Associate Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002530
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Dyssomnias
MeSH Terms: conditions — Dyssomnias | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep Application Diary (Experimental): A sleep application diary which will automatically report results back to sleep doctor is used in addition to standard sleep hygiene counseling.
  Interventions: Behavioral: Sleep Application Diary; Behavioral: Treatment As Usual
- Treatment as Usual (Active Comparator): Sleep hygiene counseling
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Sleep Application Diary — Tool used to document sleep hygiene.
  Arms: Sleep Application Diary
Behavioral: Treatment As Usual — Sleep hygiene counseling

SUMMARY:
The purpose of this study will be to see if adolescents can advance bedtime above what can be accomplished by counseling alone simply by inputting their information into a sleep application diary and reporting this information back to their sleep doctor.

DETAILED DESCRIPTION:
Using a smart phone application, participants will record bedtime and wake up times as well as answer questions about their sleep throughout their participation in this study . Reaction time will also be measured through a smart phone application.

ELIGIBILITY:
Inclusion Criteria:

* Males & Females age 12-17
* have access to a smart phone (iphone or android)
* present to a sleep disorder clinic with poor sleep hygiene and seen by a pediatric sleep specialist

Exclusion Criteria:

* significant developmental delays
* English is not the primary language spoken

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Time to Bed | 1 month, 3 months, & 6 months
  improvement in consistency of time to bed

SECONDARY OUTCOMES:
Reaction Time | 1 month, 3 months, & 6 months
  reaction time measured by reaction time test application

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Tierney, MD, MPH, Principal Investigator — Penn State College of Medicine, Milton S. Hershey Medical Center
Locations (5):
- United States (5):
  - 30 Hope Drive, Hershey, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Hershey Children's Hospital-Lancaster Outpatient, Lancaster, Pennsylvania
  - Penn State Hershey Medical Group-St. Joes, Reading, Pennsylvania
  - Penn State Hershey Medical Group-York-Apple hill, York, Pennsylvania

REFERENCES:
- [Background] Behar J, Roebuck A, Domingos JS, Gederi E, Clifford GD. A review of current sleep screening applications for smartphones. Physiol Meas. 2013 Jul;34(7):R29-46. doi: 10.1088/0967-3334/34/7/R29. Epub 2013 Jun 17. PMID 23771214
- [Background] Stippig A, Hubers U, Emerich M. Apps in sleep medicine. Sleep Breath. 2015 Mar;19(1):411-7. doi: 10.1007/s11325-014-1009-6. Epub 2014 Jun 3. PMID 24888483
- [Background] Egton Medical Information System Limited (2014). Sleep Diary Patient.co.uk (Version 1.3) [Mobile application software]. Retrieved from http://itunes.apple.com
- [Background] Lenhart, A., Ling, R., Campbell, S., Purcell, K. (2010, April 20). Teens and Mobile Phones. Pew Research Center's Internet & Amerian Life Project. Retrieved December 8, 2011 from http://www.pewinternet.org/2010/04/20/teens-and-mobile-phones/
- [Background] Shirazi, Alireza Sahami, James Clawson, Yashar Hassanpour, Mohammad J. Tourian, Albrecht Schmidt, Ed H. Chi, Marko Borazio, and Kristof Van Laerhoven.
- [Background] Bassan, Fabio. (2014). Ultra Reaction-who is faster? (Version 1.5) [Mobile application software]. Retrieved from http://itunes.apple.com
- [Background] Qiwii. (2013). Reaction time (version 1.0.0). [Mobile application software]. Retrieved from http://play.google.com